CLINICAL TRIAL: NCT03466333
Title: Feasibility Study on the Effects of Postnatal Enalapril on Maternal Cardiovascular Function Following Preterm Pre-eclampsia.
Brief Title: Postnatal Enalapril to Improve Cardiovascular fUnction Following Preterm Pre-eclampsia
Acronym: PICk-UP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R04725
Record Dates: First submitted 2018-03-08; First posted 2018-03-15 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Cardiovascular Diseases; Pre-Eclampsia Onset Less Than 37 Weeks (Diagnosis)
Keywords: preterm pre-eclampsia; cardiovascular dysfunction
MeSH Terms: conditions — Cardiovascular Diseases; Disease | interventions — Enalapril

STUDY DESIGN:
Intervention Model Description: Double blind randomised controlled trial (40 participants) Eligible women who decline to take art in the interventional arm, can consent to the observational arm of the study (up to 40 participants)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Investigational medicinal product (Experimental): Oral enalapril maleate once daily: 5mg for 1 week, then 10mg for 2 weeks, then 20mg maintenance (for total of 6 months postpartum)
  Interventions: Drug: Enalapril Maleate
- Placebo (Placebo Comparator): Oral placebo once daily for 6 months postpartum
  Interventions: Drug: Placebo oral capsule
- Observational arm (No Intervention): For participants who decline to be take part in the interventional part of the study (decline randomisation to IMP/placebo) however they consent to the observational components of the study (serial echocardiography and biomarkers postpartum).

INTERVENTIONS:
Drug: Enalapril Maleate — Enalapril maleate will be encapsulated; participants will take the drug once a day for 6 months following delivery.
  Arms: Investigational medicinal product
Drug: Placebo oral capsule — The placebo will be encapsulated; participants will take the drug once a day for 6 months following delivery. It will be identical in appearance to the IMP.
  Arms: Placebo

SUMMARY:
This is a double blind randomised controlled feasibility study investigating the effect of postnatal enalapril on cardiovascular function in women who have had preterm pre-eclampsia. Participants will be randomised to 6 months of enalapril or placebo within 3 days of delivery. Cardiovascular function will be assessed using serial echocardiography and biomarkers.

DETAILED DESCRIPTION:
Pre-eclampsia (PE) is a condition in pregnancy, identified by a combination of high blood pressure and protein in the urine. It affects 3-5% pregnancies. Women with preterm PE (pPE; delivery before 37 weeks) frequently develop abnormal heart function after pregnancy, which increases their risk of heart disease in later life. Subtle changes in heart function have also been shown to increase the chance of a woman getting PE again in her next pregnancy. Despite this, research to date has focused on the pregnancy and relatively little is known about what happens after pregnancy and whether outcomes can be improved with treatment. sFlt is a protein that prevents blood vessel growth and causes blood vessel constriction. sFlt levels are raised in pPE and correlate with the degree of abnormal heart function. In animal studies, sFlt has been shown to directly cause injury to the heart and it is therefore possible that sFlt mediates pPE associated heart damage. Angiotensin converting enzyme (ACE) inhibitors are commonly used to protect against heart damage following myocardial infarction, but their use has never been tested following pPE.

Objectives:

1. To characterise abnormal heart function following pPE
2. To determine if this can be modified by treatment with enalapril.

Study design:

Women who have had pPE, will be randomly allocated to enalapril or placebo from delivery for 6 months. Heart function will be assessed using blood tests and ultrasound scans (echocardiography). This will allow us to learn more about how pPE affects the heart (from the placebo group) and measure the protective effect of enalapril on the heart. Recruitment rates and acceptability of the intervention will also be assessed in this feasibility study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pPE in this pregnancy requiring delivery < 37 weeks gestation: new or worsening hypertension >20 weeks with proteinuria or other features suggestive of PE (abnormal haematological, biochemical parameters, fetal growth restriction (FGR) and/or abnormal sFlt:PlGF (>85)).
* Biochemical / haematological cut-offs:
* Platelet count <100 x109/L
* Alanine amino transferase > 50units/L
* Creatinine >90mmol/L
* FGR:
* Abdominal circumference (AC) / estimated fetal weight (EFW) <3rd centile
* Or 2 of the following:
* AC/EFW <10th centile
* AC/EFW crossing centiles by >2 quartiles
* Cerebroplacental ratio <5th centile
* Umbilical artery PI >95th centile
* At time of randomisation:
* Postpartum, within 3 days of delivery
* Aged 18 years or over
* Able to provide informed consent
* Serum creatinine <100 mmol/l

Exclusion Criteria:

* Inability to consent
* Known cardiac disease
* Contraindication to ACE inhibitors
* Renal artery stenosis

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
Process outcome | 24 months
  Recruitment rate (number of women eligible, recruited and completing the study per month)
Clinical outcome | 32 months
  Reduction in total vascular resistance (TVR) (from baseline to 6 months post-randomisation following treatment with enalapril, compared with placebo). Whilst TVR is the nominated primary endpoint for this feasibility study, the choice of primary outcome for the definitive trial remains uncertain.

SECONDARY OUTCOMES:
Process outcome | 32 months
  Acceptability of the intervention to postnatal women.
Clinical outcome (echocardiography measures) | 32 months
  A change in other parameters of cardiac function (including: E/E' ratio, tricuspid valve regurgitation, left atrial volume index (LAVi), left ventricular function (LVEF), cardiac output (CO), stroke volume (SV), relative wall thickness (RWT), left ventricular mass index (LVMi), concentric/eccentric remodelling, global longitudinal strain (GLS), left ventricular (LV) basal strain, LV apical strain)
Clinical outcome (biomarkers) | 32 months
  A change in biomarkers (high sensitivity troponin (hs-cTnT), placental growth factor (PlGF), soluble fms-like tyrosine kinase-1 (sFlt1), N-terminal pro-brain natriuretic peptide (NTproBNP), nitric oxide end products (NOx).

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Dr Myers, MBBS PhD, Principal Investigator — The University of Manchester
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

REFERENCES:
- [Derived] Ormesher L, Higson S, Luckie M, Roberts SA, Glossop H, Trafford A, Cottrell E, Johnstone ED, Myers JE. Postnatal Enalapril to Improve Cardiovascular Function Following Preterm Preeclampsia (PICk-UP):: A Randomized Double-Blind Placebo-Controlled Feasibility Trial. Hypertension. 2020 Dec;76(6):1828-1837. doi: 10.1161/HYPERTENSIONAHA.120.15875. Epub 2020 Oct 5. PMID 33012200